CLINICAL TRIAL: NCT03024970
Title: Daily Disposable Dispensing Clinical Trial of Test Lens Against Stenfilcon A Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-16-60
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- stenfilcon A lens with solution additive (test) (Experimental): Participants were randomized to wear the stenfilcon A lens with solution additive (test) for 1 month during the cross over study.
  Interventions: Device: stenfilcon A lens with solution additive (test); Device: stenfilcon A lens (control)
- stenfilcon A lens (control) (Active Comparator): Participants were randomized to wear stenfilcon A (control) lens pair for 1 month during the cross over study.
  Interventions: Device: stenfilcon A lens with solution additive (test); Device: stenfilcon A lens (control)

INTERVENTIONS:
Device: stenfilcon A lens with solution additive (test) — silicone hydrogel lens
Device: stenfilcon A lens (control) — contact lens

SUMMARY:
The purpose of this study is to investigate the overall clinical performance of the test daily disposable stenfilcon A lens with solution additive (test) compared to the stenfilcon A lens (control).

DETAILED DESCRIPTION:
This will be, prospective, multicenter, double-masked, randomized, bilateral, 1 month cross-over, dispensing study comparing the test lens against the stenfilcon A control lens with a study duration of approximately two months.

Each subject will be randomized to wear either the test or control as a matched pair first and subjects will be randomized based on the order in which the subject is enrolled and qualified into the study.

ELIGIBILITY:
Inclusion Criteria:

* A person is eligible for inclusion in the study if he/she:

  * Has had a self-reported oculo-visual examination in the last two years.
  * Is at least 18 years of age and has full legal capacity to volunteer.
  * Has read and understood the information consent letter.
  * Is willing and able to follow instructions and maintain the appointment schedule.
  * Is correctable to a visual acuity of 20/40 or better (in each eye) with their habitual vision correction or 20/20 best-corrected.
  * Must achieve 20/30 or better (in each eye) with study lenses
  * Requires spectacle lens powers between -0.75 and -6.50 diopters sphere (0.25D steps).
  * Has no more than 0.75 diopters of refractive astigmatism.
  * Currently wears soft contact lenses.
  * Have clear corneas and no active ocular disease.
  * Has not worn lenses for at least 12 hours before the examination

Exclusion Criteria:

* A person will be excluded from the study if he/she:

  * Has never worn contact lenses before.
  * Has any systemic disease affecting ocular health.
  * Is using any systemic or topical medications that will affect ocular health.
  * Has any ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses.
  * Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
  * Has any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars.
  * Is aphakic.
  * Has undergone corneal refractive surgery.
  * Is pregnant, lactating, or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit).
  * Have taken part in any other contact lens or care solution clinical trial or research, within one week prior to starting this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-01; Primary Completion 2017-04-25 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pete Kollbaum, OD, PhD, Principal Investigator — Clinical Optics Research Lab (CORL) Indiana University School of Optometry.; Eric Ritchey, OD, PhD, FAAO, Principal Investigator — University of Houston
Locations (2):
- United States (2):
  - Clinical Optical Research Lab (CORL), Bloomington, Indiana
  - The Ocular Surface Institute (TOSI), Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Lens Then Control Lens: Participants were randomized to wear the stenfilcon A lens with solution additive (test) for 1 month during the cross over study.
  stenfilcon A lens with solution additive (test): contact lens stenfilcon A lens (Control): contact lens
- Control Lens Then Test Lens: Participants were randomized to wear stenfilcon A (control) lens pair for 1 month during the cross over study.
  stenfilcon A lens (control): contact lens stenfilcon A lens with solution additive (test): contact lens
Period: First Intervention
Arm/Group | Test Lens Then Control Lens | Control Lens Then Test Lens
Started | 34 | 38
Completed | 33 | 38
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Second Intervention
Arm/Group | Test Lens Then Control Lens | Control Lens Then Test Lens
Started | 33 | 38
Completed | 32 | 38
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 72
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Subjective Ratings on Comfort
Description: Subjects assessed comfort for test and control lens on a scale 0-10, 0=not comfortable 10=comfortable
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
units on a scale | 9.7 (0.6) | 9.6 (0.7)

2. Primary Outcome: Subjective Ratings on Comfort
Description: Subjects assessed comfort for test and control lens on a scale 0-10, 0=not comfortable 10=comfortable
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
units on a scale | 9.1 (1.5) | 9.0 (1.5)

3. Primary Outcome: Subjective Ratings on Comfort
Description: Subjects assessed comfort for test and control lens on a scale 0-10, 0=not comfortable 10=comfortable
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
units on a scale | 8.9 (1.7) | 8.6 (1.9)

4. Primary Outcome: Vision Satisfaction
Description: Subjective ratings on vision satisfaction was assessed for test and control lens using a 5- point Likert scale: 1- Strongly disagree, 2- disagree, 3- neutral, 4- agree, 5- strongly agree
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
percentage of participants
  Strongly disagree | 0 | 0
  Disagree | 0 | 0
  Neutral | 6 | 1
  Agree | 39 | 39
  Strongly agree | 55 | 60

5. Primary Outcome: Vision Satisfaction
Description: as for outcome 4
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
percentage of participants
  Strongly disagree | 0 | 1
  Disagree | 3 | 1
  Neutral | 3 | 4
  Agree | 29 | 26
  Strongly agree | 65 | 68

6. Primary Outcome: Vision Satisfaction
Description: as for outcome 4
Time Frame: 1 Month
Measure: Number; unit: percentage of participants
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
percentage of participants
  Strongly disagree | 3 | 1
  Disagree | 1 | 3
  Neutral | 4 | 9
  Agree | 34 | 26
  Strongly agree | 58 | 61

7. Primary Outcome: Visual Acuity On High Illumination High Contrast
Description: Visual acuity is assessed on high illumination high contrast logMAR charts for test and control lenses. Visual acuity of logMar of 0.0 is equivalent to 20/20 of Snellen. Each 0.1 addition in logMar is 1 line in Snellen chart.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
LogMAR | -0.20 (0.06) | -0.21 (0.06)

8. Primary Outcome: Visual Acuity On High Illumination High Contrast
Description: Visual acuity is assessed on high illumination high contrast for test and control lens by LogMAR. Visual acuity of logMar of 0.0 is equivalent to 20/20 of Snellen. Each 0.1 addition in logMar is 1 line in Snellen chart.
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
LogMAR | -0.21 (0.06) | -0.20 (0.06)

9. Primary Outcome: Visual Acuity On High Illumination High Contrast
Description: as for outcome 8
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
LogMAR | -0.21 (0.07) | -0.20 (0.05)

10. Primary Outcome: Visual Acuity On Low Illumination High Contrast
Description: Visual acuity is assessed on low illumination high contrast for test and control lens by LogMAR. Visual acuity of logMar of 0.0 is equivalent to 20/20 of Snellen. Each 0.1 addition in logMar is 1 line in Snellen chart.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
LogMAR | -0.08 (0.09) | -0.09 (0.09)

11. Primary Outcome: Visual Acuity On Low Illumination High Contrast
Description: as for outcome 10
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
LogMAR | -0.09 (0.10) | -0.09 (0.09)

12. Primary Outcome: Visual Acuity On Low Illumination High Contrast
Description: as for outcome 10
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
LogMAR | -0.09 (0.10) | -0.09 (0.09)

13. Primary Outcome: Overall Corneal Staining
Description: Overall corneal staining is assessed for test and control lens in a scale of 0-4, 0=No staining,1=trace, 2=mild, 3=moderate, 4=Severe.
Time Frame: One Week
Measure: Number; unit: percentage of participants
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
percentage of participants
  Grade 0 | 55 | 57
  Garde 1 | 31 | 27
  Grade 2 | 14 | 14
  Grade 3 | 0 | 2
  Grade 4 | 0 | 0

14. Primary Outcome: Overall Corneal Staining
Description: as for outcome 13
Time Frame: One Month
Measure: Number; unit: percentage of participants
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
percentage of participants
  Grade 0 | 54 | 58
  Garde 1 | 33 | 30
  Grade 2 | 13 | 11
  Grade 3 | 0 | 1
  Grade 4 | 0 | 0

15. Primary Outcome: Conjunctival Staining
Description: Conjunctival staining is assessed for test and control lens in 0.50 steps. Scale 0-4, 0=None, 4= Deep confluent
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 0.36 (0.45) | 0.39 (0.43)

16. Primary Outcome: Conjunctival Staining
Description: Conjunctival staining is assessed for test and control lens in 0.50 steps. Scale 0-4, 0=None, 4= Deep confluent
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 0.42 (0.37) | 0.45 (0.43)

17. Primary Outcome: Bulbar Hyperemia
Description: Bulbar hyperemia is assessed for test and control lens on a scale of 0-4,0.25 steps. (0=None, 1=Slight injection of conjunctival vessels, 2=Mild injection, 3=Moderate injection, 4=Severe injection)
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 1.32 (0.85) | 1.28 (0.78)

18. Primary Outcome: Bulbar Hyperemia
Description: as for outcome 17
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 1.36 (0.81) | 1.33 (0.82)

19. Primary Outcome: Limbal Hyperemia
Description: Limbal hyperemia is assessed for test and control lens on a scale of 0-4,0.25 steps. (0=None, 1=Slight injection of conjunctival vessels, 2=Mild injection, 3=Moderate injection, 4=Severe injection)
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 0.85 (0.64) | 0.89 (0.68)

20. Primary Outcome: Limbal Hyperemia
Description: as for outcome 19
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 0.90 (0.66) | 0.78 (0.67)

21. Primary Outcome: Palpebral Hyperemia
Description: Palpebral hyperemia is assessed for test and control lens on a scale of 0-4,0.25 steps. (0=None, 1=Slight injection of conjunctival vessels, 2=Mild injection, 3=Moderate injection, 4=Severe injection)
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 0.89 (0.65) | 0.88 (0.63)

22. Primary Outcome: Palpebral Hyperemia
Description: as for outcome 21
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 1.02 (0.63) | 0.93 (0.55)

23. Secondary Outcome: Lens Fit Acceptance
Description: Overall fit acceptance is assessed for test and control lens. Scale 0-4, 0=can't be worn, 1=Poor, 2=Fair, 3=Good, 4=optimum.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 3.4 (0.3) | 3.3 (0.3)

24. Secondary Outcome: Lens Fit Acceptance
Description: as for outcome 23
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 3.3 (0.3) | 3.3 (0.3)

25. Secondary Outcome: Lens Fit Acceptance
Description: as for outcome 23
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 3.3 (0.3) | 3.2 (0.5)

26. Secondary Outcome: Handling Satisfaction
Description: Handling satisfaction is assessed for test and control lens. 5 point Likert scale: 1- Strongly disagree, 2-disagree, 3-neutral, 4-agree, 5- strongly agree
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
percentage of participants
  Strongly disagree | 0 | 0
  Disagree | 0 | 1
  Neutral | 3 | 1
  Agree | 25 | 23
  Strongly Agree | 72 | 75

27. Secondary Outcome: Handling Satisfaction
Description: as for outcome 26
Time Frame: 1 Month
Measure: Number; unit: percentage of participants
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
percentage of participants
  Strongly disagree | 0 | 1
  Disagree | 0 | 4
  Neutral | 1 | 0
  Agree | 30 | 23
  Strongly Agree | 69 | 72

28. Secondary Outcome: Lens Surface - Wettability
Description: Wettability is assessed for test and control lens on a scale of 0-4, 0=Very poor, 4=Excellent
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 3.52 (0.36) | 3.52 (0.35)

29. Secondary Outcome: Lens Surface - Wettability
Description: Wettability is assessed for test and control lens on a scale of 0-4, 0=Very poor, 4=Excellent
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 3.47 (0.46) | 3.33 (0.48)

30. Secondary Outcome: Lens Surface - Wettability
Description: Wettability is assessed for test and control lens on a scale of 0-4, 0=Very poor, 4=Excellent
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 3.37 (0.43) | 3.38 (0.44)

31. Secondary Outcome: Lens Surface - Deposits
Description: Deposits are assessed for test and control lens. Scale 0-4, 0.25 steps. 0=Clean, no deposits, 4=Deposits of 0.5mm or larger or film covering more than 75% of surface.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 0.03 (0.15) | 0.02 (0.15)

32. Secondary Outcome: Lens Surface - Deposits
Description: as for outcome 31
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 0.04 (0.20) | 0.04 (0.19)

33. Secondary Outcome: Lens Surface - Deposits
Description: as for outcome 31
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
Number analyzed (Eyes) | 140 | 140
units on a scale | 0.06 (0.27) | 0.02 (0.15)

34. Secondary Outcome: Subjective Ratings on Dryness
Description: Subjective ratings on dryness is assessed for test and control lens on a scale of 0-10, 0=dry, 10=not dry
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
units on a scale | 9.6 (1.3) | 9.5 (0.9)

35. Secondary Outcome: Subjective Ratings on Dryness
Description: Subjective ratings on dryness is assessed for test and control lens on a scale of 0-10, 0=dry, 10=not dry
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
units on a scale | 8.8 (1.8) | 8.8 (1.6)

36. Secondary Outcome: Subjective Ratings on Dryness
Description: Subjective ratings on dryness is assessed for test and control lens on a scale of 0-10, 0=dry, 10=not dry
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
Number analyzed (Participants) | 70 | 70
units on a scale | 8.3 (2.1) | 8.1 (2.3)

ADVERSE EVENTS:
Time Frame: From baseline up to 1 month on each pair of lenses.
Arm/Group | Stenfilcon A Lens With Solution Additive (Test) | Stenfilcon A Lens (Control)
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 1/72 | 5/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stenfilcon A Lens With Solution Additive (Test) (N=72) | Stenfilcon A Lens (Control) (N=72)
Corneal Staining (Eye disorders) | 1 (1) | 2 (2)
Subconjuctival Hyperemia (Eye disorders) | 0 (0) | 2 (2)
Epithelial defect (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/70/NCT03024970/Prot_SAP_000.pdf